CLINICAL TRIAL: NCT05957393
Title: Improving Physician Vaccine Recommendation Using Social Norms, Trust, and Presumptive Language
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: Pro00113696
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2023-10

CONDITIONS: Healthy
Keywords: Physicians; Vaccination Recommendation; Social Norms; Trust; Presumptive Recommendation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Quantity (present) x Quality (present) (Experimental): Participants will receive a social norm-based message (for quantity) and will learn the AIMS method, a trust-building method using presumptive language (for quality).
  Interventions: Other: Quantity of vaccination recommendations; Other: Quality of vaccination recommendations
- Quantity (present) x Quality (absent) (Experimental): Participants will receive a social norm-based message (for quantity).
  Interventions: Other: Quantity of vaccination recommendations
- Quantity (absent) x Quality (present) (Experimental): Participants will learn the AIMS method, a trust-building method using presumptive language (for quality).
  Interventions: Other: Quality of vaccination recommendations
- Quantity (absent) x Quality (absent) (Experimental): Control: Participants in this condition will receive general information about vaccines, including vaccine principles, uptake barriers, and guidelines. This information will come directly from the CDC's Advisory Committee on Immunization Practices (ACIP) website.
  Interventions: Other: Control

INTERVENTIONS:
Other: Quantity of vaccination recommendations — The survey contains a messaging intervention using a 2x2 randomized factorial design, where the investigators attempt to increase the quantity and/or quality of physician and APP vaccination recommendations (Quantity (present vs. absent) x Quality (present vs. absent)).
  Arms: Quantity (present) x Quality (absent); Quantity (present) x Quality (present)
Other: Quality of vaccination recommendations — The survey contains a messaging intervention using a 2x2 randomized factorial design, where the investigators attempt to increase the quantity and/or quality of physician and APP vaccination recommendations (Quantity (present vs. absent) x Quality (present vs. absent)).
  Arms: Quantity (absent) x Quality (present); Quantity (present) x Quality (present)
Other: Control — The survey contains a messaging intervention using a 2x2 randomized factorial design, where the investigators attempt to increase the quantity and/or quality of physician and APP vaccination recommendations (Quantity (present vs. absent) x Quality (present vs. absent)).
  Arms: Quantity (absent) x Quality (absent)

SUMMARY:
This research examines vaccination recommendation perceptions and behaviors of physicians and advanced practice providers.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be physicians, advanced practice providers, medical students, nurses/nurse practitioners, or medical fellows.
* Must be in a position to be authorized to recommend vaccines to patients in their official professional capacities/responsibilities.

Exclusion Criteria:

* Students or employees under the supervision of the PI who meet inclusion criteria for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Change in proportion of patients that receive a vaccine recommendation | Day 1, Day 30, Day 60, Day 90
  Proportion of patients that receive a vaccine recommendation = multiplication of the answer to the following two items: (1) "I (will) check(ed) whether a patient has/had gotten all indicated vaccines", (2) "If I saw/see a patient had not gotten an indicated vaccine, I (will) discuss(ed) getting it." Both items are answered on a scale from 0% (never) to 100% (always).
Change in self-reported responsibility perception | Day 1, Day 30, Day 60, Day 90
  Self-reported responsibility perception = answer to the following item: (1) "Recommending indicated vaccines is within the scope of my professional responsibilities". This item is answered on a scale from 0% (completely disagree) to 100% (completely agree).
Change in self-reported assessment of patient recommendation acceptance | Day 1, Day 30, Day 60, Day 90
  Self-reported assessment of patient recommendation acceptance = answer to the following item: (1) "If I recommend(ed) an indicated vaccine, my patient (will) accept(ed) that recommendation.". This item is answered on a scale from 0% (never) to 100% (always).
Change in self-reported patient trust | Day 1, Day 30, Day 60, Day 90
  Self-reported patient trust = answer to the following item: (1) "Thinking about the last/next 30 days I provided care, I can say that my patients (will) trust(ed) me as their healthcare provider". This item is answered on a scale from 0% (completely disagree) to 100% (completely agree).
Change in self-reported utilization of AIMS | Day 1, Day 30, Day 60, Day 90
  Composite score of the following items: (1) "I used/will use direct, declarative language, like: "You're due for your flu shot. We'll do that at the end of this visit"; (2) "If the patient showed/shows hesitancy about getting vaccinated, I (will) ask(ed) about their concerns, and then use(d) active listening to understand their thoughts"; (3) "If the patient showed/shows hesitancy about getting vaccinated, I (will) listen(ed) to the patient's reasoning and then summarize(d) the patient's reasoning back to them to show that I understood/understand"; (4) "If the patient still has concerns, I did/will not continue efforts to convince them."
  Each item is answered on a scale from 0% (never) to 100% (always).
Change in self-reported rate of patient vaccine uptake | Day 1, Day 30, Day 60, Day 90
  Answer to the following item: "Estimate what percentage of your patients is/will be fully vaccinated against […]" This item is answered on a scale from 0% to 100%.
  The question is being asked 8-10 times with the following name inserted for [...] in the above question:
  Flu COVID-19 Tetanus, Diphtheria, Pertussis HPV Hepatitis B Meningitis / Meningococcal Shingles Pneumococcal Other (which can be two other diseases that the respondent indicated)

SECONDARY OUTCOMES:
Change in belief about patient autonomy | Day 1, Day 30, Day 60, Day 90
  Answer to the following item: "I stated / will state the patient's options - to vaccinate or not, and with which vaccine - so that they can make an informed decision." This item is answered on a scale from 0% to 100%.
Change in proportion of patients that accept a recommendation | Day 1, Day 30, Day 60, Day 90
  Proportion of patients that accept a recommendation = multiplication of the answer to the following three items: (1) "I (will) check(ed) whether a patient has/had gotten all indicated vaccines", (2) "If I saw/see a patient had not gotten an indicated vaccine, I (will) discuss(ed) getting it."; (3) "If I recommend(ed) an indicated vaccine, my patient (will) accept(ed) that recommendation." All items are answered on a scale from 0% (never) to 100% (always).

CONTACTS AND LOCATIONS:
Overall Officials: Dan Ariely, PhD, Principal Investigator — Duke University
Locations (3):
- United States (2):
  - (Any and all facilities) - The study team ask(s)/(ed) professional contacts, friends, and family members who are employed at various US Institutions to forward the recruitment announcement message via their respective networks, Durham, North Carolina
  - Duke University Health System (all locations), Durham, North Carolina
- (Any and all facilities) - Participants are recruited via market research company "Survey Healthcare Global", Brasília, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Personal information will be permanently removed from the data no later than two weeks after the distribution of the final study survey, after which study responses will no longer be able to be linked to an individual participant.
  What specific individual participant data sets are to be shared: Answers to all questions in all surveys will be shared.
Supporting Information: SAP
Time Frame: After data from the last participant is collected, we'll take 6 months for analysis before data becomes available. Data will be available indefinitely.
Access Criteria: Disaggregated data will be uploaded to the Open Science Framework research portal.